CLINICAL TRIAL: NCT06802588
Title: Optimization of the Management of Non-Traumatic Intracerebral Hemorrhage (OPT-ICH)
Acronym: OPT-ICH
Status: Recruiting | Type: Observational
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Other Study IDs: 2022_011
Record Dates: First submitted 2025-01-07; First posted 2025-01-31 (Actual); Last update posted 2026-01-15 (Actual); Status verified 2026-01

CONDITIONS: Intracerebral Hemorrhage
MeSH Terms: conditions — Cerebral Hemorrhage

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — routine blood samples
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Intracerebral non-traumatic intraparenchymal hemorrhages (ICH) account for 15 to 20% of strokes. One third of the patients dies within the month following ICH, and survivors often experience residual disability with a high risk of recurrent ICH, other serious vascular events, and neurological complications such as epilepsy and dementia. Encouraging but preliminary data suggest a favorable trend in terms of survival rates in recent years. This is partly due to improved management of patients with ICH, which must be early (the concept of "time is brain") and carried out by expert personnel (medical and paramedical) in specialized units.

The main objectives of the study are:

* To evaluate the management of patients with ICH in the acute phase within the University Hospital of Tours by analyzing the procedures adopted in the various relevant departments (neurovascular units, neurosurgery, medical or neurosurgical intensive care, geriatrics);
* To evaluate whether the systematic implementation of a dedicated protocol (see *) for the management of patients with ICH is associated with a reduction in mortality and disability in the short and long term.

DETAILED DESCRIPTION:
The project consists of 2 parts:

* Retrospective, multicentric, observational study. Inclusion of all patients presenting with ICH admitted urgently to the University Hospital of Tours between 2018-2021.
* Prospective, multicentric, observational study. Inclusion of all patients presenting with ICH admitted urgently to the University Hospital of Tours, Angers and Poitiers.

Each patient will benefit from management according to a protocol which will include:

* Emergency MRI with contrast injection (contrast-enhanced brain CT scan if contraindicated);
* Admission to the Neurovascular Unit unless hemodynamically unstable or intubated;
* First intravenous antihypertensive injection with a goal < 1 hour from arrival at the hospital;
* Anticoagulation reversal with a goal < 1 hour from arrival at the hospital;
* Standard laboratory tests + coagulation study ;
* Neurosurgical consultation upon arrival at the department;
* Follow-up MRI at 24-48 hours or earlier if clinical worsening;
* Diagnostic work-up for the evaluation of hypertension-related end organ damage (Transthoracic echocardiogram, retinography , proteinuria);
* Contrast-enhanced follow-up MRI at 3-6 months;
* Neurological evaluation at 6 months and 2 years;
* When applicable a neuropsychological evaluation at 6M and 2 Y;

ELIGIBILITY:
Inclusion Criteria:

* aged over 18 years
* emergency admission to the University Hospital of Tours
* having an ICH on imaging performed upon admission (CT scan or MRI) at the University Hospital of Tours

Exclusion criteria :

- Patient who has given their opposition to the collection of their data

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult population with acute ICH
Sampling Method: Probability Sample
Enrollment: 600 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
mortality and disability | 6 months, 2 years
  Primary Outcome Measure Title:
  Modified Rankin Scale (mRS) Scores to Assess Disability and Mortality
  Description:
  The study will evaluate functional outcomes, disability, and mortality in patients with non-traumatic intracerebral hemorrhage. Functional outcomes will be measured using the modified Rankin Scale (mRS), which evaluates the degree of disability or dependence in daily activities. The mRS scores range from 0 (no symptoms) to 6 (death). Data will be summarized as the proportion of participants in each mRS category at 6 months and 2 years. Mortality will be assessed as the percentage of participants with an mRS score of 6.

SECONDARY OUTCOMES:
Neuropsychiatric patient profile among the survivors | 6 months, 2 years
  Cognitive and behavioral outcomes will be measured using a battery of neuropsychiatric tests, including assessments for memory, executive function, attention, and mood disorders (e.g., depression and anxiety). Data will be reported as mean test scores for each domain

CONTACTS AND LOCATIONS:
Overall Officials: Marco PASI, MD, PHD, Principal Investigator — neurovascular unit, neurology department, CHRU Tours; Grégoire Boulouis, MD, PHD, Principal Investigator — interventionnal neuroradiology unit, neuroradiology department, CHRU Tours
Locations (3):
- France (3):
  - University Hospital of Angers, Angers
  - University Hospital of Poitiers, Poitiers
  - University Hospital Center of Tours, Tours

IPD SHARING:
Plan to Share IPD: No